CLINICAL TRIAL: NCT05126108
Title: Evaluation of the Decurarisation Kinetics of Rocuronium in Cervical Surgery
Brief Title: Decurarisation Kinetics of Rocuronium in Cervical Surgery
Acronym: CIDEROC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210278
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Non-morbidly Obese Patients (BMI<35); Equiring General Anesthesia With Intubation With a Nerve Integrity Monitor (NIM) Tube; Thyroid and Parathyroid Surgery
Keywords: Thyroid and parathyroid surgery; Recurrent nerves monitoring; Rocuronium
MeSH Terms: conditions — Thyroid Diseases | interventions — Thyroid (USP)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Thyroid and parathyroid surgery — Thyroid and parathyroid surgery
Other: Recurrent nerves monitoring — Recurrent nerves monitoring

SUMMARY:
Recurrent nerve monitoring for thyroid and parathyroid surgery contraindicates the pharmacologically active presence of muscle relaxant agents at the time of dissection. A recent formalized expert guideline (RFE 2018) from the French Society of Anesthesia and Resuscitation, SFAR recommends administering a curare to facilitate tracheal intubation and limit laryngeal trauma . This study aims to determine if the level of neuromuscular recovery is consistent with monitoring the recurrent nerve after the use of rocuronium for intubation.

Primary endpoint: Achievement of quality intraoperative laryngeal recurrent nerve monitoring.

DETAILED DESCRIPTION:
The monitoring of the recurrent nerves, innervating the vocal cords, in thyroid and parathyroid surgery has developed in recent years because of its interest as a parameter to reduce the risk of recurrent paralysis.

Monitoring of the recurrent nerves requires contraction of the laryngeal muscle and therefore contraindicates the pharmacologically active presence of muscle relaxants at the time of dissection. Thus, intubation was performed either without curare or with a depolarizing curare (Succinylcholine) whose short duration of action allowed optimal intubation conditions without intraoperative residual effect.

This practice is being questioned due to :

(i) a recent formalized expert referential (RFE) of the French Society of Anesthesia and Resuscitation, SFAR, which recommends administering a curare to facilitate intubation of the trachea and limit laryngeal trauma (grade 1 +) and (ii) a restriction of the indications of succinylcholine by the French National Agency for the Safety of Medicines and Health Products, ANSM, as an adjuvant of general anaesthesia (induction in rapid sequence and electroconvulsive therapy).

In summary, thyroid surgery requires curarisation for intubation and sufficient intraoperative decurarisation to allow monitoring of the recurrent nerves. We hypothesize that the time between intubation and the actual start of recurrent monitoring is consistent with the time to recovery of laryngeal adductor neuromuscular block after injection of rocuronium at a dosage of 0.5 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects requiring general anesthesia for cephalic surgery (thyroid and parathyroid) with an NIM-type intubation tube.
* Subject informed of the study and not having opposed it

Exclusion Criteria:

* Allergy to any of the products used
* Morbidly obese subjects (BMI> 35)
* Pregnancy
* Predictive criteria for difficult intubation in pre-anesthetic consultation
* Subjects under tutorship or curatorship
* Subjects not affiliated to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major, non-morbidly obese patients (BMI<35) requiring general anesthesia with intubation with a Nerve Integrity Monitor (NIM) tube for thyroid and parathyroid surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Quality intraoperative monitoring of the recurrent laryngeal nerve | During surgery
  To assess the decurarization kinetics of rocuronium: to determine if the level of neuromuscular recovery is compatible with monitoring of the recurrent nerve after the use of rocuronium for intubation

SECONDARY OUTCOMES:
Copenhagen score | During surgery
  Evaluate the intubation conditions 3 minutes after the injection of rocuronium
Arterial pressions | During surgery
  Evaluate the hemodynamic variations induced by anesthetic induction
Cardiac frequency | During surgery
  Evaluate the hemodynamic variations induced by anesthetic induction

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical anesthesia service - Cochin Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marquet Y, Philippe A, Toussaint S, Abdallah SB, Morel-Fatio E, Baillard C. Rocuronium with sugammadex as a rescue reversal agent to solve conflicting recommendations for thyroid or parathyroid surgery. A prospective study. Anaesth Crit Care Pain Med. 2023 Aug;42(4):101214. doi: 10.1016/j.accpm.2023.101214. Epub 2023 Mar 6. PMID 36889437